CLINICAL TRIAL: NCT04122729
Title: Study of the N680S Polymorphism of the FSHR Gene and Its Relationship With the Type of Gonadotropin Used in Controlled Ovarian Stimulation
Brief Title: N680S Polymorphism of the FSHR Gene and Its Relationship With the Type of Gonadotropin Used in COS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Angelini Farmacéutica (Industry)
Collaborators: Sistemas Genómicos (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANG-FOS-2019-01
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: In Vitro Fertilization; Controlled Ovarian Stimulation
Keywords: Highly purified human follicle stimulating hormone (HP-FSH); Recombinant follicle stimulating hormone (rFSH); FSH receptor (FSHR); Polymorphism N680S of the FSHR; Polymorphism N312S of the LHCGR; LHCG receptor (LHCGR); Polymorphism c.2039G>A; Polymorphism c.935A>G

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood samples suitable for molecular analysis and DNA samples extraction. Once the determinations are made, these blood samples will be destroyed.
Oversight: Data Monitoring Committee: No

SUMMARY:
This project wants to determinate whether there is a relationship between the N680S polymorphism genotype of the FSHR gene and the nature of the FSH used in controlled ovarian stimulation.

It is a non-interventional, observational, cross-sectional and retrospective, national and multicenter study, in which a genetic test will be carried out to determine the genotype of the N680S polymorphism in samples of blood of patients who have undergone two cycles of controlled ovarian stimulation in the last 8 months.

DETAILED DESCRIPTION:
The investigators want to investigate whether the N680S polymorphism of the FSRH gene could affects ovarian response with different nature of the FSH used (human FSH and recombinant FSH) in patients undergoing two consecutive cycles of IVF/ICSI with controlled ovarian stimulation.

All patients who agree to participate in the study will have a blood sample taken on the same day as a routine extraction performed for the 2nd cycle of the controlled ovarian stimulation in accordance with the standard clinical practice of each hospital. The sample will be sent to the central laboratory to determine the genotype of the afore mentioned polymorphism and correlate it with the clinical results obtained with the two cycles of controlled ovarian stimulation.

In order to avoid any bias, the study population will follow a crossover design with respect to the type of FSH used in the first and second cycles of the COS (i.e., half of the recruited patients must have undergone a first cycle of COS with recombinant FSH and a second cycle with human FSH; and, conversely, the other half must have undergone a first cycle with human FSH and a second cycle with recombinant FSH). In order to avoid potential modifications to the inclusion criteria, the time elapsed between the two cycles should not exceed 6 months.

ELIGIBILITY:
Inclusion criteria:

* Signature of Informed Consent
* Age ≤ 37 years
* BMI < 30 kg/m2
* Antral follicles count 1st cycle COS = 5-15
* Antimüllerian hormone basal 1st cycle COS > 1,1 ng/ml and < 3,1 ng/ml
* COS protocol: equal starting dose in the 2 cycles of COS (150-225 UI/day) with dose adjustment from the 5th day of COS; pituitary suppression protocol in the 2 cycles of COS with GnRH antagonist with onset when ≥ 1 follicle of ≥ 14 mm in diameter or E2 ≤ 600 pg/ml; and triggering with hCGr or GnRH agonist
* Optional the use of oral contraceptives (OC) (however, same in the 2 cycles)
* 4-9 recovered oocytes in the 1st cycle of COS
* ≤ 6 months between the 2 cycles of COS

Exclusion criteria:

* Use of the LH activity during the cycles of COS
* Presence of severe male factor
* Grade III-IV endometriosis
* Patients with polycystic ovary syndrome, a history of uterine or ovarian surgeries, hydrosalpinx visible by ultrasound, or uterine fibroids measuring > 30 mm
* Major systemic or uncontrolled endocrine-metabolic diseases affecting the pituitary gland, the thyroid gland, the adrenal glands, the pancreas, the liver, or the kidneys

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing two cycles of IVF/ICSI who achieved a suboptimal response after the 1st cycle, did not become pregnant, and consequently underwent another cycle of COS in which the protocol was amended during the 2nd cycle to change the nature of the FSH used during the 1st cycle.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Oocytes retrieved | Through study completion, an average of 1 year
  Number of oocytes retrieved in each IVF/ICSI cycle with controlled ovarian stimulation used different nature of the FSH in each one (human FSH and recombinant FSH).
Genotype of the N680S polymorphism of the FSHR gene | Through study completion, an average of 1 year
  Genotype of the N680S polymorphism of the FSHR gene will be tested on blood samples

SECONDARY OUTCOMES:
Genotype of the N312S polymorphism of the LHCGR gene | Through study completion, an average of 1 year
  Genotype of the N312S polymorphism of the LHCGR gene will be tested on blood samples

CONTACTS AND LOCATIONS:
Overall Officials: María Carrera, PhD, Study Director — Hospital Universitario 12 de Octubre
Locations (12):
- Spain (12):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Clínic, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Virgen de las Nieves, Granada
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trounson AO, Leeton JF, Wood C, Webb J, Wood J. Pregnancies in humans by fertilization in vitro and embryo transfer in the controlled ovulatory cycle. Science. 1981 May 8;212(4495):681-2. doi: 10.1126/science.7221557. PMID 7221556
- [Background] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332
- [Background] Kligman I, Rosenwaks Z. Differentiating clinical profiles: predicting good responders, poor responders, and hyperresponders. Fertil Steril. 2001 Dec;76(6):1185-90. doi: 10.1016/s0015-0282(01)02893-x. PMID 11730748
- [Background] Freour T, Masson D, Mirallie S, Jean M, Bach K, Dejoie T, Barriere P. Active smoking compromises IVF outcome and affects ovarian reserve. Reprod Biomed Online. 2008 Jan;16(1):96-102. doi: 10.1016/s1472-6483(10)60561-5. PMID 18252054
- [Background] Coccia ME, Rizzello F. Ovarian reserve. Ann N Y Acad Sci. 2008 Apr;1127:27-30. doi: 10.1196/annals.1434.011. PMID 18443326
- [Background] Broekmans FJ, Kwee J, Hendriks DJ, Mol BW, Lambalk CB. A systematic review of tests predicting ovarian reserve and IVF outcome. Hum Reprod Update. 2006 Nov-Dec;12(6):685-718. doi: 10.1093/humupd/dml034. Epub 2006 Aug 4. PMID 16891297
- [Background] Broer SL, Broekmans FJ, Laven JS, Fauser BC. Anti-Mullerian hormone: ovarian reserve testing and its potential clinical implications. Hum Reprod Update. 2014 Sep-Oct;20(5):688-701. doi: 10.1093/humupd/dmu020. Epub 2014 May 12. PMID 24821925
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Polyzos NP, Nwoye M, Corona R, Blockeel C, Stoop D, Haentjens P, Camus M, Tournaye H. Live birth rates in Bologna poor responders treated with ovarian stimulation for IVF/ICSI. Reprod Biomed Online. 2014 Apr;28(4):469-74. doi: 10.1016/j.rbmo.2013.11.010. Epub 2013 Dec 4. PMID 24581984
- [Background] Sunkara SK, Coomarasamy A, Faris R, Braude P, Khalaf Y. Long gonadotropin-releasing hormone agonist versus short agonist versus antagonist regimens in poor responders undergoing in vitro fertilization: a randomized controlled trial. Fertil Steril. 2014 Jan;101(1):147-53. doi: 10.1016/j.fertnstert.2013.09.035. Epub 2013 Nov 1. PMID 24188873
- [Background] Steward RG, Lan L, Shah AA, Yeh JS, Price TM, Goldfarb JM, Muasher SJ. Oocyte number as a predictor for ovarian hyperstimulation syndrome and live birth: an analysis of 256,381 in vitro fertilization cycles. Fertil Steril. 2014 Apr;101(4):967-73. doi: 10.1016/j.fertnstert.2013.12.026. Epub 2014 Jan 23. PMID 24462057
- [Background] van Loendersloot LL, van Wely M, Limpens J, Bossuyt PM, Repping S, van der Veen F. Predictive factors in in vitro fertilization (IVF): a systematic review and meta-analysis. Hum Reprod Update. 2010 Nov-Dec;16(6):577-89. doi: 10.1093/humupd/dmq015. Epub 2010 Jun 25. PMID 20581128
- [Background] van der Gaast MH, Eijkemans MJ, van der Net JB, de Boer EJ, Burger CW, van Leeuwen FE, Fauser BC, Macklon NS. Optimum number of oocytes for a successful first IVF treatment cycle. Reprod Biomed Online. 2006 Oct;13(4):476-80. doi: 10.1016/s1472-6483(10)60633-5. PMID 17007663
- [Background] Verberg MF, Eijkemans MJ, Macklon NS, Heijnen EM, Baart EB, Hohmann FP, Fauser BC, Broekmans FJ. The clinical significance of the retrieval of a low number of oocytes following mild ovarian stimulation for IVF: a meta-analysis. Hum Reprod Update. 2009 Jan-Feb;15(1):5-12. doi: 10.1093/humupd/dmn053. PMID 19091754
- [Background] Polyzos NP, Sunkara SK. Sub-optimal responders following controlled ovarian stimulation: an overlooked group? Hum Reprod. 2015 Sep;30(9):2005-8. doi: 10.1093/humrep/dev149. Epub 2015 Jul 21. PMID 26202582
- [Background] Cascorbi I, Bruhn O, Werk AN. Challenges in pharmacogenetics. Eur J Clin Pharmacol. 2013 May;69 Suppl 1:17-23. doi: 10.1007/s00228-013-1492-x. Epub 2013 May 3. PMID 23640184
- [Background] Altmae S, Hovatta O, Stavreus-Evers A, Salumets A. Genetic predictors of controlled ovarian hyperstimulation: where do we stand today? Hum Reprod Update. 2011 Nov-Dec;17(6):813-28. doi: 10.1093/humupd/dmr034. Epub 2011 Aug 23. PMID 21862569
- [Background] Overbeek A, Lambalk N. Pharmacogenomics of ovulation induction: facilitating decisions on who, when and how to treat. Pharmacogenomics. 2009 Sep;10(9):1377-9. doi: 10.2217/pgs.09.110. No abstract available. PMID 19761360
- [Background] Loutradis D, Theofanakis C, Anagnostou E, Mavrogianni D, Partsinevelos GA. Genetic profile of SNP(s) and ovulation induction. Curr Pharm Biotechnol. 2012 Mar;13(3):417-25. doi: 10.2174/138920112799361954. PMID 21657995
- [Background] Gromoll J, Ried T, Holtgreve-Grez H, Nieschlag E, Gudermann T. Localization of the human FSH receptor to chromosome 2 p21 using a genomic probe comprising exon 10. J Mol Endocrinol. 1994 Jun;12(3):265-71. doi: 10.1677/jme.0.0120265. PMID 7916967
- [Background] Simoni M, Gromoll J, Nieschlag E. The follicle-stimulating hormone receptor: biochemistry, molecular biology, physiology, and pathophysiology. Endocr Rev. 1997 Dec;18(6):739-73. doi: 10.1210/edrv.18.6.0320. No abstract available. PMID 9408742
- [Background] Aittomaki K, Lucena JL, Pakarinen P, Sistonen P, Tapanainen J, Gromoll J, Kaskikari R, Sankila EM, Lehvaslaiho H, Engel AR, Nieschlag E, Huhtaniemi I, de la Chapelle A. Mutation in the follicle-stimulating hormone receptor gene causes hereditary hypergonadotropic ovarian failure. Cell. 1995 Sep 22;82(6):959-68. doi: 10.1016/0092-8674(95)90275-9. PMID 7553856
- [Background] Yao Y, Ma CH, Tang HL, Hu YF. Influence of follicle-stimulating hormone receptor (FSHR) Ser680Asn polymorphism on ovarian function and in-vitro fertilization outcome: a meta-analysis. Mol Genet Metab. 2011 Aug;103(4):388-93. doi: 10.1016/j.ymgme.2011.04.005. Epub 2011 Apr 17. PMID 21546300
- [Background] Laan M, Grigorova M, Huhtaniemi IT. Pharmacogenetics of follicle-stimulating hormone action. Curr Opin Endocrinol Diabetes Obes. 2012 Jun;19(3):220-7. doi: 10.1097/MED.0b013e3283534b11. PMID 22499219
- [Background] Huang X, Li L, Hong L, Zhou W, Shi H, Zhang H, Zhang Z, Sun X, Du J. The Ser680Asn polymorphism in the follicle-stimulating hormone receptor gene is associated with the ovarian response in controlled ovarian hyperstimulation. Clin Endocrinol (Oxf). 2015 Apr;82(4):577-83. doi: 10.1111/cen.12573. Epub 2014 Oct 3. PMID 25132286
- [Background] Perez Mayorga M, Gromoll J, Behre HM, Gassner C, Nieschlag E, Simoni M. Ovarian response to follicle-stimulating hormone (FSH) stimulation depends on the FSH receptor genotype. J Clin Endocrinol Metab. 2000 Sep;85(9):3365-9. doi: 10.1210/jcem.85.9.6789. PMID 10999835
- [Background] Lledo B, Guerrero J, Turienzo A, Ortiz JA, Morales R, Ten J, Llacer J, Bernabeu R. Effect of follicle-stimulating hormone receptor N680S polymorphism on the efficacy of follicle-stimulating hormone stimulation on donor ovarian response. Pharmacogenet Genomics. 2013 May;23(5):262-8. doi: 10.1097/FPC.0b013e32835fe813. PMID 23470615
- [Background] van Wely M, Kwan I, Burt AL, Thomas J, Vail A, Van der Veen F, Al-Inany HG. Recombinant versus urinary gonadotrophin for ovarian stimulation in assisted reproductive technology cycles. Cochrane Database Syst Rev. 2011 Feb 16;2011(2):CD005354. doi: 10.1002/14651858.CD005354.pub2. PMID 21328276
- [Background] Lledo B, Dapena P, Ortiz JA, Morales R, Llacer J, Bernabeu R. Clinical efficacy of recombinant versus highly purified follicle-stimulating hormone according to follicle-stimulating hormone receptor genotype. Pharmacogenet Genomics. 2016 Jun;26(6):288-93. doi: 10.1097/FPC.0000000000000215. PMID 26959715
- [Background] Ascoli M, Fanelli F, Segaloff DL. The lutropin/choriogonadotropin receptor, a 2002 perspective. Endocr Rev. 2002 Apr;23(2):141-74. doi: 10.1210/edrv.23.2.0462. PMID 11943741
- [Background] Puett D, Li Y, DeMars G, Angelova K, Fanelli F. A functional transmembrane complex: the luteinizing hormone receptor with bound ligand and G protein. Mol Cell Endocrinol. 2007 Jan 2;260-262:126-36. doi: 10.1016/j.mce.2006.05.009. Epub 2006 Oct 23. PMID 17059864
- [Background] Rousseau-Merck MF, Misrahi M, Atger M, Loosfelt H, Milgrom E, Berger R. Localization of the human luteinizing hormone/choriogonadotropin receptor gene (LHCGR) to chromosome 2p21. Cytogenet Cell Genet. 1990;54(1-2):77-9. doi: 10.1159/000132962. PMID 2249480
- [Background] Rousseau-Merck MF, Atger M, Loosfelt H, Milgrom E, Berger R. The chromosomal localization of the human follicle-stimulating hormone receptor gene (FSHR) on 2p21-p16 is similar to that of the luteinizing hormone receptor gene. Genomics. 1993 Jan;15(1):222-4. doi: 10.1006/geno.1993.1041. PMID 8432542
- [Background] Fanelli F, Puett D. Structural aspects of luteinizing hormone receptor: information from molecular modeling and mutagenesis. Endocrine. 2002 Aug;18(3):285-93. doi: 10.1385/ENDO:18:3:285. PMID 12450321
- [Background] Fanelli F, Themmen AP, Puett D. Lutropin receptor function: insights from natural, engineered, and computer-simulated mutations. IUBMB Life. 2001 Mar;51(3):149-55. doi: 10.1080/152165401753544214. PMID 11547916
- [Background] Capalbo A, Sagnella F, Apa R, Fulghesu AM, Lanzone A, Morciano A, Farcomeni A, Gangale MF, Moro F, Martinez D, Ciardulli A, Palla C, Uras ML, Spettu F, Cappai A, Carcassi C, Neri G, Tiziano FD. The 312N variant of the luteinizing hormone/choriogonadotropin receptor gene (LHCGR) confers up to 2.7-fold increased risk of polycystic ovary syndrome in a Sardinian population. Clin Endocrinol (Oxf). 2012 Jul;77(1):113-9. doi: 10.1111/j.1365-2265.2012.04372.x. PMID 22356187
- [Background] Lindgren I, Baath M, Uvebrant K, Dejmek A, Kjaer L, Henic E, Bungum M, Bungum L, Cilio C, Leijonhufvud I, Skouby S, Andersen CY, Giwercman YL. Combined assessment of polymorphisms in the LHCGR and FSHR genes predict chance of pregnancy after in vitro fertilization. Hum Reprod. 2016 Mar;31(3):672-83. doi: 10.1093/humrep/dev342. Epub 2016 Jan 14. PMID 26769719
- [Background] Valkenburg O, Uitterlinden AG, Piersma D, Hofman A, Themmen AP, de Jong FH, Fauser BC, Laven JS. Genetic polymorphisms of GnRH and gonadotrophic hormone receptors affect the phenotype of polycystic ovary syndrome. Hum Reprod. 2009 Aug;24(8):2014-22. doi: 10.1093/humrep/dep113. Epub 2009 Apr 29. PMID 19403562
- [Background] Piersma D, Verhoef-Post M, Look MP, Uitterlinden AG, Pols HA, Berns EM, Themmen AP. Polymorphic variations in exon 10 of the luteinizing hormone receptor: functional consequences and associations with breast cancer. Mol Cell Endocrinol. 2007 Sep 30;276(1-2):63-70. doi: 10.1016/j.mce.2007.06.007. Epub 2007 Jul 17. PMID 17709176
- [Background] Simoni M, Tuttelmann F, Michel C, Bockenfeld Y, Nieschlag E, Gromoll J. Polymorphisms of the luteinizing hormone/chorionic gonadotropin receptor gene: association with maldescended testes and male infertility. Pharmacogenet Genomics. 2008 Mar;18(3):193-200. doi: 10.1097/FPC.0b013e3282f4e98c. PMID 18300940